CLINICAL TRIAL: NCT02944435
Title: A Comparative, Randomized, Single-Dose, 2-Way Crossover Pharmacokinetic Comparability Study of CB-839 Administered as Capsule and Tablet Formulations in Healthy Adult Subjects
Brief Title: A Comparative, Pharmacokinetic Study of CB-839 Capsule and Tablet Formulations in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CX-839-006
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Healthy Volunteers
Keywords: Glutaminase Inhibitor; Glutaminase; CB-839
MeSH Terms: interventions — CB-839

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CB-839 Capsules (Experimental): A single dose of 3 x 200-mg capsules of CB-839 will be administered orally with water approximately 5 minutes after consuming an entire meal
  Interventions: Drug: CB-839 Capsules
- CB-839 Tablets (Active Comparator): A single dose of 3 x 200-mg tablets of CB-839 will be administered orally with water approximately 5 minutes after consuming an entire meal
  Interventions: Drug: CB-839 Tablets

INTERVENTIONS:
Drug: CB-839 Capsules — 3 x 200 mg CB-839 Capsules (Reference Formulation)
  Other Names: Glutaminase inhibitor
  Arms: CB-839 Capsules
Drug: CB-839 Tablets — 3 x 200 mg CB-839 Tablets (Test Formulation)
  Other Names: Glutaminase inhibitor
  Arms: CB-839 Tablets

SUMMARY:
This is a Phase 1, randomized, single-dose, 2-way crossover PK comparability study of CB-839 administered as capsule and tablet formulations in healthy adult subjects.

DETAILED DESCRIPTION:
A new tablet formulation of CB-839 was recently developed in order to enable rapid, automated manufacturing of CB-839. Previous studies have used a capsule formulation of CB-839. This study will enable a PK comparison between CB-839 capsules and CB-839 tablets.

This is a Phase 1, comparative, randomized, single-dose, 2-way crossover PK comparability study of CB-839 administered as capsule and tablet formulations in healthy adult subjects. Serial blood samples for PK analyses will be collected over a 24 hour period after each administration of CB-839. All subjects will be monitored for safety throughout their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, 18-55 years of age, inclusive, at screening.
* Has not used nicotine containing products for at least 3 mo prior the first dose.
* Body mass index (BMI) within 18.0 and 30.0 kg/m2, inclusively, at screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECGs, as deemed by the Principal Investigator (PI).
* For a female of childbearing potential: either be sexually inactive (abstinent) for 14 days prior to the first dose and through 14 days following the last dose of study drug(s) or be using one of the following acceptable birth control methods:

  1. Non-hormone releasing intrauterine device in place for at least 3 mo prior to the first dose of study drug with either a physical (e.g., condom, diaphragm) or a chemical (e.g., spermicide) barrier method from the time of screening through 14 days following the last dose of study drug.
  2. A physical barrier method (e.g., condom, diaphragm) with a chemical barrier method (e.g., spermicide) for at least 14 days prior to the first dose of study drug and until 14 days after the last dose of study drug.
* In addition, female subjects of childbearing potential will be advised to remain sexually inactive or to keep the same birth control method or for at least 14 days following the last dose of study drug.
* For a female of non-childbearing potential: must have undergone one of the following sterilization procedures at least 6 mo prior to the first dose of study drug:

  1. hysteroscopic sterilization;
  2. bilateral tubal ligation or bilateral salpingectomy;
  3. non-surgical transcervical sterilization (e.g., Essure®);
  4. hysterectomy;
  5. bilateral oophorectomy;
  6. or be postmenopausal with amenorrhea for at least 1 year prior to the first CB-839 dose with FSH serum levels consistent with postmenopausal status as per PI judgment.
* A non-vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 mo or more prior to study start. A male who has been vasectomized less than 4 mo prior to study start must follow the same restrictions as a non-vasectomized male).
* If male, must agree not to donate sperm from dosing until 90 days after the last dose.
* Understands the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol.

Exclusion Criteria:

* Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or is expected to manifest significant emotional problems during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI.
* History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* History or presence of alcoholism or drug abuse within the past 2 years prior to screening.
* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or inactive ingredient(s).
* History or presence of:

  1. liver disease, pancreatic insufficiency or intestinal malabsorption;
  2. neuropathy or muscle disorders;
  3. seizures;
  4. asthma;
  5. fluid retention;
  6. cardiovascular disease, cardiac arrhythmias, hypertension, cardiovascular thrombotic events, myocardial infarction, or stroke;
  7. ulcer disease or gastrointestinal bleeding;
  8. renal papillary necrosis and other renal injury;
  9. exfoliative dermatitis, Stevens-Johnson syndrome, and toxic epidermal necrolysis.
* Female subjects who are pregnant or lactating.
* Positive urine drug or alcohol results at screening or check-in.
* Positive urine cotinine at screening.
* Positive results at screening for HIV types 1 and 2, HBsAg, or HCV.
* Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
* Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
* QTcF interval is > 460 msec (males) or > 480 msec (females) or deemed clinically abnormal by the PI at screening.
* Estimated creatinine clearance < 90 mL/min at screening.
* Unable to refrain from or anticipates the use of:

  1. Any non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dose of study drug and throughout the study.
  2. Any prescription medications (including hormonal contraceptives, hormone replacement therapy, and lithium) beginning 14 days prior to the first dose of study drug and throughout the study.
  3. Proton pump inhibitors (PPIs) beginning 14 days prior to the first dose of study drug and throughout the study.
* Has been on a diet incompatible with the on-study diet (in the opinion of the PI) within the 28 days prior to the first dose of study drug, and throughout the study.
* Donation of blood or significant blood loss within 56 days prior to the first dose of study drug.
* Plasma donation within 14 days prior to the first dose of study drug.
* Participation in another clinical trial within 28 days prior to the first dose of study drug. The 28-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Comparison of Area Under the Curve (AUC) of CB-839 capsules and CB-839 tablets | -0.5 hr (predose), 0.5, 1, 2, 4, 5, 6, 8, 10, 12 and 24 hours postdose on Day 1 & Day 3
  To compare the AUC from time zero to the last measurable concentration and from zero to infinity of a single 600 mg dose of CB-839 tablets (Test) and a single 600 mg dose of CB-839 capsules (Reference Treatment)
Comparison of Maximum Concentrations (Cmax) of CB-839 capsules and CB-839 tablets | -0.5 hr (predose), 0.5, 1, 2, 4, 5, 6, 8, 10, 12 and 24 hours postdose on Day 1 & Day 3
  To compare the Cmax of a single 600 mg dose of CB-839 tablets (Test) and a single 600 mg dose of CB-839 capsules (Reference Treatment)
Comparison of Time to Observed Maximum Concentrations (Tmax) of CB-839 capsules and CB-839 tablets | -0.5 hr (predose), 0.5, 1, 2, 4, 5, 6, 8, 10, 12 and 24 hours postdose on Day 1 & Day 3
  To compare the Tmax of a single 600 mg dose of CB-839 tablets (Test) and a single 600 mg dose of CB-839 capsules (Reference Treatment)
Comparison of the Apparent Terminal Elimination Half-Life of CB-839 capsules and CB-839 tablets | -0.5 hr (predose), 0.5, 1, 2, 4, 5, 6, 8, 10, 12 and 24 hours postdose on Day 1 & Day 3
  To compare the apparent terminal elimination half-life of a single 600 mg dose of CB-839 tablets (Test) and a single 600 mg dose of CB-839 capsules (Reference Treatment)
Comparison of the Apparent Terminal Elimination Rate Constant of CB-839 capsules and CB-839 tablets | -0.5 hr (predose), 0.5, 1, 2, 4, 5, 6, 8, 10, 12 and 24 hours postdose on Day 1 & Day 3
  To compare the apparent terminal elimination rate constant of a single 600 mg dose of CB-839 tablets (Test) and a single 600 mg dose of CB-839 capsules (Reference Treatment)
The safety of CB-839 capsules and tablets by examining incidence, severity, relationship, type of AE, changes in clinical laboratory tests (hematology, serum chemistry, urinalysis), physical examination, 12-lead ECGs, vital signs and concomitant therapy | 8 days
  Subjects will be monitored for safety by examining the incidence, severity, relationship, and type of AE as well as changes in clinical laboratory tests (hematology, serum chemistry, urinalysis), physical examination, 12-lead ECGs, vital signs and concomitant therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Peterson, MD, Principal Investigator — Algorithme Pharma USA LLC
Locations (1):
- Algorithme Pharma USA, LLC, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No